CLINICAL TRIAL: NCT00417937
Title: A Multicenter, Double-Blind Clinical Trial to Assess the Efficacy and Tolerability of Topical Azelaic Acid 15% Gel Once Daily Compared to Topical Azelaic Acid 15% gelTwice Daily in Subjects With Papulopustular Rosacea
Brief Title: A Multicenter Trial of a Topical Medication for Papulopustular Rosacea Applied Twice Daily Versus Once Daily
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14428; 1401460 (Other: Company internal)
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2014-02

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Azelaic acid 15 % gel once daily
  Interventions: Drug: azelaic acid 15% gel
- 2 (Active Comparator): Azelaic acid 15 gel twice daily
  Interventions: Drug: azelaic acid 15% gel

INTERVENTIONS:
Drug: azelaic acid 15% gel — 15% gel, topically applied once daily for six weeks
  Arms: 1
Drug: azelaic acid 15% gel — 15% gel, topically applied twice daily for six weeks
  Arms: 2

SUMMARY:
To assess the efficacy and tolerability of azelaic acid 15% gel applied once daily versus twice daily in the treatment of patients with papulopustular rosacea.

DETAILED DESCRIPTION:
To test the efficacy and safety of once vs twice daily application of azelaic acid 15% gel on papulopustular rosacea

ELIGIBILITY:
Inclusion Criteria:

- Papulopustular facial rosacea; minimum of 10, maximum of 50 inflamed papules and/or pustules

Exclusion Criteria:

* Mild or severe rosacea
* Rosacea with marked ocular manifestations
* Presence of dermatoses that could interfere with the rosacea diagnosis or evaluation of the study course
* Wash out period required for patients treated prior to study with topical retinoids, oral antibiotics, topical antibiotics, systemic and topical corticosteroids, topical imidazole, laser surgery for telangiectasia
* History of hypersensitivity to propylene glycol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Investigator's global assessment scored on a seven point scale | Measurements made during the course of treatment

SECONDARY OUTCOMES:
Inflammatory lesion count, erythema, telangiectasia, patient self assessment, patient opinion about therapy | Parameters measured during the course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Intendis GmbH, Berlin, Germany